CLINICAL TRIAL: NCT00081939
Title: A Phase 2 Study Incorporating Bone Marrow Microenvironment (ME) Co-Targeting Bortezomib Into Tandem Melphalan-Based Autotransplants With DT PACE for Induction/Consolidation and Thalidomide + Dexamethasone for Maintenance
Brief Title: UARK 2003-33, Total Therapy III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2003-33
Record Dates: First submitted 2004-04-27; First posted 2004-04-29 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Treatment (Experimental): Two cycles of VDTPACE induction (Velcade days 1, 4, 8, and 11; DTPACE days 4-7) with interim thalidomide (50 mg QD) + Dex (20 mg QD x 4 days every 21 days) following each cycle. Induction followed by single or tandem MEL200 transplant (MEL140 mg/m2 for subjects > 70 years of age) with interim thalidomide (100mg QD) + Dex (20 mg QD x 4 days every 21 days) following each transplant. Transplants followed by two cycles of VDTPACE consolidation (Velcade days 1, 4, 8, and 11; DTPACE days 1-4) with interim thalidomide (100mg QD) + Dex (20 mg QD x 4 days every 21 days) following each cycle of VDTPACE. Consolidation followed by 3 years of maintenance therapy with VDT (velcade 1.0 mg/m2 days 1, 4, 8, 11 q 28 days; Thal 100 mg QD; and Dex 20mg days 1-4 and 8-11 q 28 days) during Year 1 and TD (Thal 100 mg QD and Dex 20 mg days 1-4, q 28 days) or VTD (velcade 1.0 mg/m2 weekly, Thal 100 mg QD, and Dex 20 mg weekly) during Years 2 and 3.
  Interventions: Drug: Velcade; Drug: Thalidomide

INTERVENTIONS:
Drug: Velcade — Two cycles of induction on days 1,4,8,11 at 1.0mg/m^2. Two cycles of consolidation on days 1,4,8,11 at 1.0mg/m^2. Maintenance year one 1.0mg/m^2 1,4,8,11 q 28 days.
Drug: Thalidomide — Two cycles of VDTPACE 200mg thal days 4-7(cycle 1)and days 1-4 cycle 2 interim Thal 50mg qd between VTDPACE cycles and between cycle 2 and transplant. Thal 100mg between transplants d/c 7 days prior to each transplant. Consolidation therapy cycles 3 and 4 VDTPACE 200mg days 1-4 both cycles. Interim maintenance to maintenance 100mg qd. Maintenance year 1 thal 100mg qd. Maintenance years 2 and 3 Thal 100mg qd.

SUMMARY:
There have been two previous Total Therapy studies for multiple myeloma (MM) at the Myeloma Institute for Research and Therapy (MIRT): Total Therapy I (from 1989 through 1994) and Total Therapy II (from 1996 to 2004). Results have shown that patients treated on these studies had better outcomes (meaning patients have lived longer and had better responses to treatment) when compared to patients treated with standard chemotherapy.

With this new study, Total Therapy III, researchers will take what they have learned from the first two studies and add new treatment strategies to try to improve the outcomes even more, especially for patients with chromosome abnormalities.

DETAILED DESCRIPTION:
1.1 To determine, in a historical comparison with TT II (Thalidomide arm), whether two cycles of VDTPACE induction (instead of four induction cycles in TT II) followed by more timely MEL 200-based transplant with DEX + THAL between transplants can:

1.1.1 Increase the CR frequency from 50% to 60% at 18 months from initiation of therapy;

1.1.2 Increase > n-CR rate pre-transplant #1 from 20% to 40%;

1.1.3 Raise 2-year EFS rates from 55% to 75% in patients with CA and from 80% to 95%, in patients without CA.

ELIGIBILITY:
Induction Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Protein criteria must be present (quantifiable M-component of IgG, IgA, IgD, or IgE and/or urinary kappa or lambda light chain or Bence Jones protein) in order to evaluate response. Non-secretory patients are eligible provided the patient has > 20% plasmacytosis or multiple (>3) focal plasmacytomas on MRI or diffuse hyperintense signal on STIR images in the absence of hematopoietic growth factors.
* Patients must have received no more than one cycle of prior chemotherapy for this disease. Patients may have received prior radiotherapy provided approval has been obtained by the Principal Investigator.
* Patients must be < or = 75 years of age at the time of initial registration.
* Ejection fraction by ECHO or MUGA >40% performed within 60 days prior to registration.
* Patients must have adequate pulmonary function studies > or = 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > or =50% of predicted, within 60 days of registration. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, there must be a pulmonary consult documenting that the patient is a candidate for high dose therapy.
* Patients must have a performance status of 0-2 based on SWOG criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* All patients must be informed of the investigational nature of this study and must have signed an IRB-approved informed consent in accordance with institutional and federal guidelines.

Induction Exclusion Criteria:

* Platelet count < 30 x 10^9/L, unless myeloma-related
* ANC < 1.0 X 10^9/L, unless myeloma-related
* Grade > or =2 peripheral neuropathy
* Hypersensitivity to bortezomib, boron, or mannitol
* Uncontrolled diabetes.
* Recent (< or =6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
* Evidence of chronic obstructive or chronic restrictive pulmonary disease.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Pregnant or nursing women. Women of child-bearing potential must have a negative pregnancy test documented within one week of registration. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2004-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Al Hadidi S, Ababneh OE, Schinke CD, Thanendrarajan S, Siegel ER, Bailey C, Smith R, Panozzo SB, Zangari M, Tricot G, Shaughnessy JD Jr, Zhan F, Sawyer J, Barlogie B, van Rhee F. Long-Term Follow-Up of Patients With Multiple Myeloma Treated on Earlier Total Therapy Protocols: A Secondary Analysis of 3 Clinical Trials. JAMA Oncol. 2025 Aug 1;11(8):910-915. doi: 10.1001/jamaoncol.2025.1394. PMID 40471585
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481
- [Derived] Vatsveen TK, Sponaas AM, Tian E, Zhang Q, Misund K, Sundan A, Borset M, Waage A, Brede G. Erythropoietin (EPO)-receptor signaling induces cell death of primary myeloma cells in vitro. J Hematol Oncol. 2016 Aug 31;9(1):75. doi: 10.1186/s13045-016-0306-x. PMID 27581518
- [Derived] Usmani SZ, Sawyer J, Rosenthal A, Cottler-Fox M, Epstein J, Yaccoby S, Sexton R, Hoering A, Singh Z, Heuck CJ, Waheed S, Chauhan N, Johann D, Abdallah AO, Muzaffar J, Petty N, Bailey C, Crowley J, van Rhee F, Barlogie B. Risk factors for MDS and acute leukemia following total therapy 2 and 3 for multiple myeloma. Blood. 2013 Jun 6;121(23):4753-7. doi: 10.1182/blood-2012-11-466961. Epub 2013 Apr 19. PMID 23603914
- [Derived] Usmani SZ, Mitchell A, Waheed S, Crowley J, Hoering A, Petty N, Brown T, Bartel T, Anaissie E, van Rhee F, Barlogie B. Prognostic implications of serial 18-fluoro-deoxyglucose emission tomography in multiple myeloma treated with total therapy 3. Blood. 2013 Mar 7;121(10):1819-23. doi: 10.1182/blood-2012-08-451690. Epub 2013 Jan 10. PMID 23305732
- [Derived] Waheed S, Mitchell A, Usmani S, Epstein J, Yaccoby S, Nair B, van Hemert R, Angtuaco E, Brown T, Bartel T, McDonald J, Anaissie E, van Rhee F, Crowley J, Barlogie B. Standard and novel imaging methods for multiple myeloma: correlates with prognostic laboratory variables including gene expression profiling data. Haematologica. 2013 Jan;98(1):71-8. doi: 10.3324/haematol.2012.066555. Epub 2012 Jun 24. PMID 22733020
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675
- [Derived] Usmani SZ, Sexton R, Hoering A, Heuck CJ, Nair B, Waheed S, Al Sayed Y, Chauhan N, Ahmad N, Atrash S, Petty N, van Rhee F, Crowley J, Barlogie B. Second malignancies in total therapy 2 and 3 for newly diagnosed multiple myeloma: influence of thalidomide and lenalidomide during maintenance. Blood. 2012 Aug 23;120(8):1597-600. doi: 10.1182/blood-2012-04-421883. Epub 2012 Jun 6. PMID 22674807
- See also: Click here for more information about UAMS — http://www.myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Treatment
Started | 303
Completed | 303
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 219
  >=65 years | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival (PFS) at 3 Years From Initiation of Study Treatment
Description: In patients with no confirmed Partial Response, Near Complete Response, or Complete Response, progression was defined as a >25% increase from baseline in myeloma protein production or other signs of disease progression such as hypercalcemia, etc.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 303
percentage of participants | 77

ADVERSE EVENTS:
Arm/Group | Study Treatment
Serious Adverse Events (participants affected / at risk) | 303/303
Other Adverse Events (participants affected / at risk) | 303/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=303)
Grade 3 Allergic reaction/hypersensitivity (Immune system disorders) | 7
Grade 4 Allergic reaction/Hypersensitivity (Immune system disorders) | 2
Grade 4 Allergy-other (Immune system disorders) | 1
Grade 3 Autoimmune reaction (Immune system disorders) | 1
Grade 3 Hearing (Ear and labyrinth disorders) | 4
Grade 3 Anemia (HGB) (Blood and lymphatic system disorders) | 139
Grade 4 Anemia (HGB) (Blood and lymphatic system disorders) | 48
Grade 3 CD4 count (Blood and lymphatic system disorders) | 1
Grade 3 Lymphopenia (Blood and lymphatic system disorders) | 1
Grade 3 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 4
Grade 4 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 115
Grade 3 Thrombocytopenia (PLT) (Blood and lymphatic system disorders) | 6
Grade 4 Thrombocytopenia (PLT) (Blood and lymphatic system disorders) | 296
Grade 4 Leukopenia (Blood and lymphatic system disorders) | 303
Grade 3 AV Block-Type 2 (Cardiac disorders) | 1
Grade 5 Asystole (Cardiac disorders) | 1
Grade 3 Febrile Neutropenia (Cardiac disorders) | 1
Grade 3 Hypertension (Cardiac disorders) | 2
Grade 3 Hypotension (Cardiac disorders) | 4
Grade 4 Hypotension (Cardiac disorders) | 1
Grade 3 Left vent. systolic dysfunction (Cardiac disorders) | 1
Grade 4 Left vent systolic dysfunction (Cardiac disorders) | 1
Grade 3 Supra Arrhythmia: atrial fib. (Cardiac disorders) | 7
Grade 4 Supra Arrhyth: Atrial Fib (Cardiac disorders) | 1
Grade 3 Supra Arrhyth: Atrial Flut (Cardiac disorders) | 1
Grade 3 Supra Arrhyth: Sinus Brady (Cardiac disorders) | 1
Grade 4 Valvular heart disease (Cardiac disorders) | 1
Grade 3 Vasovagal episode (Cardiac disorders) | 2
Grade 5 Vent arrhyth: Bigeminy (Cardiac disorders) | 1
Grade 3 Ventricular Arrythmia (Cardiac disorders) | 7
Grade 4 Ventricular Arrythmia (Cardiac disorders) | 2
Grade 5 Ventricular Arrythmia (Cardiac disorders) | 1
Grade 3 Cardiac General (Cardiac disorders) | 2
Grade 3 Cardiac ischemia/infarction (Cardiac disorders) | 3
Grade 4 Cardiac ischemia/infarction (Cardiac disorders) | 3
Grade 4 Cardiopulmonary arrest (Cardiac disorders) | 1
Grade 3 Hypertension (Cardiac disorders) | 4
Grade 3 Coagulation-other (Blood and lymphatic system disorders) | 1
Grade 3 Constitutional symptoms-other (General disorders) | 6
Grade 4 Constitutional symptoms-other (General disorders) | 1
Grade 5 Constitutional symptoms-other (General disorders) | 1
Grade 3 Fatigue-lethargy, malaise, asthenia (General disorders) | 157
Grade 4 Fatigue-lethargy, malaise, asthenia (General disorders) | 36
Grade 3 Fatigue-malaise, lethargy (General disorders) | 1
Grade 3 Fever (in absence of neutropenia) (General disorders) | 4
Grade 5 Fever (absence of neutropenia) (General disorders) | 1
Grade 3 Insomnia (General disorders) | 3
Grade 4 Insomnia (General disorders) | 1
Grade 3 Obesity (General disorders) | 1
Grade 3 Sweating (General disorders) | 1
Grade 3 Weight loss (General disorders) | 1
Grade 3 Weight gain (General disorders) | 1
Grade 3 Dermatology-other (Skin and subcutaneous tissue disorders) | 1
Grade 3 Dry skin (Skin and subcutaneous tissue disorders) | 1
Grade 3 Pruritus (Skin and subcutaneous tissue disorders) | 2
Grade 3 Skin rash/desquamation (Skin and subcutaneous tissue disorders) | 21
Grade 4 Skin rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Grade 3 Ulceration (Skin and subcutaneous tissue disorders) | 2
Grade 3 Diabetes (Endocrine disorders) | 12
Grade 3 Hot flashes (Endocrine disorders) | 1
Grade 3 Anorexia (Gastrointestinal disorders) | 107
Grade 4 Anorexia (Gastrointestinal disorders) | 5
Grade 3 Colitis (Gastrointestinal disorders) | 26
Grade 4 Colitis (Gastrointestinal disorders) | 3
Grade 5 Colitis (Gastrointestinal disorders) | 2
Grade 3 Constipation (Gastrointestinal disorders) | 10
Grade 4 Constipation (Gastrointestinal disorders) | 2
Grade 3 Dehydration (Gastrointestinal disorders) | 12
Grade 3 Diarrhea (Gastrointestinal disorders) | 76
Grade 4 Diarrhea (Gastrointestinal disorders) | 3
Grade 3 Distension (Gastrointestinal disorders) | 2
Grade 3 Dry mouth (Gastrointestinal disorders) | 2
Grade 3 Dysphagia (Gastrointestinal disorders) | 25
Grade 3 Esophagitis (Gastrointestinal disorders) | 22
Grade 3 GI Necrosis gallblader (Gastrointestinal disorders) | 1
Grade 3 GI Obstruction cecum (Gastrointestinal disorders) | 1
Grade 4 GI Obstruction cecum (Gastrointestinal disorders) | 1
Grade 3 GI Perforation appendix (Gastrointestinal disorders) | 2
Grade 3 GI-other (Gastrointestinal disorders) | 6
Grade 3 Gastritis (Gastrointestinal disorders) | 1
Grade 3 Heartburn (Gastrointestinal disorders) | 1
Grade 3 Hemorrhoids (Gastrointestinal disorders) | 2
Grade 3 Mucositis/Stomatitis (Gastrointestinal disorders) | 28
Grade 4 Mucositis/Stomatitis (Gastrointestinal disorders) | 3
Grade 3 Nausea (Gastrointestinal disorders) | 56
Grade 4 Nausea (Gastrointestinal disorders) | 1
Grade 3 Taste alteration (Gastrointestinal disorders) | 1
Grade 3 Vomiting (Gastrointestinal disorders) | 18
Grade 4 Vomiting (Gastrointestinal disorders) | 1
Grade 3 Hematoma (Blood and lymphatic system disorders) | 1
Grade 3 Hemorrhage, lower GI (Blood and lymphatic system disorders) | 1
Grade 4 Hemorrhage, lower GI (Blood and lymphatic system disorders) | 1
Grade 3 Hemorrhage, upper GI (Blood and lymphatic system disorders) | 3
Grade 3 Hemorrhage-other (Blood and lymphatic system disorders) | 1
Grade 3 Alkaline phosphatase increase (Hepatobiliary disorders) | 8
Grade 3 Bilirubin increase (Hepatobiliary disorders) | 12
Grade 4 Bilirubin increase (Hepatobiliary disorders) | 12
Grade 4 Bilirubin increase (Hepatobiliary disorders) | 1
Grade 3 Cholecystitis (Hepatobiliary disorders) | 1
Grade 3 Hypoalbuminemia (Hepatobiliary disorders) | 53
Grade 3 SGOT (AST) increase (Hepatobiliary disorders) | 14
Grade 4 SGOT (AST) increase (Hepatobiliary disorders) | 3
Grade 3 SGPT (ALT) increase (Hepatobiliary disorders) | 18
Grade 4 SGPT (ALT) increase (Hepatobiliary disorders) | 3
Grade 3 Colitis infectious (Infections and infestations) | 12
Grade 4 Colitis infectious (Infections and infestations) | 2
Grade 3 Febrile neutropenia (Infections and infestations) | 1
Grade 3 Febrile neutropenia (ANC, fever) (Infections and infestations) | 103
Grade 4 Febrile neutropenia (ANC, fever) (Infections and infestations) | 3
Grade 3 GI Infection 3-4 ANC abdomen (Infections and infestations) | 4
Grade 3 GI Infection 3-4 ANC Appendix (Infections and infestations) | 2
Grade 3 GI Infection 3-4 ANC Colon (Infections and infestations) | 1
Grade 3 GI Infection Unk ANC Abdomen (Infections and infestations) | 1
Grade 3 GU Infection 3-4 ANC Bladder (Infections and infestations) | 3
Grade 3 GU Infection Unk ANC UTI (Infections and infestations) | 1
Grade 3 Infection 3-4 ANC Blood (Infections and infestations) | 11
Grade 4 Infection 3-4 ANC Blood (Infections and infestations) | 1
Grade 3 Infection 3-4 ANC Cath-related (Infections and infestations) | 3
Grade 3 Infection 3-4 ANC Wound (Infections and infestations) | 1
Grade 3 Infection Unk ANC Cath-related (Infections and infestations) | 1
Grade 3 Infection Unk ANC for body (Infections and infestations) | 1
Grade 3 Infection (documented clinically or microbiologically) (Infections and infestations) | 29
Grade 3 Infection w/normal ANC Musculoskeletal (Infections and infestations) | 1
Grade 3 Infection w/normal ANC skin (Infections and infestations) | 1
Grade 3 Infection w/normal ANC GI mild (Infections and infestations) | 2
Grade 3 Infection w/normal ANC Dermatology (Infections and infestations) | 1
Grade 3 Infection w/normal ANC Gastrointestinal (Infections and infestations) | 1
Grade 3 Infection w/normal ANC General (Infections and infestations) | 7
Grade 3 Infection w/normal ANC Neurology (Infections and infestations) | 1
Grade 3 Infection w/normal ANC Renal/Genitourinary (Infections and infestations) | 1
Grade 3 Infection w/unknown ANC (Infections and infestations) | 1
Grade 5 Infection w/unknown ANC (Infections and infestations) | 1
Grade 3 Infection Clinical Doc. w/high ANC/Pulmonary (Infections and infestations) | 2
Grade 3 Infection Normal ANC Lung (Bronchus) (Infections and infestations) | 28
Grade 3 Infection Normal Lung (Pneumonia) (Infections and infestations) | 5
Grade 3 Infection other (Infections and infestations) | 1
Grade 3 Lung infection-Bronchus (Infections and infestations) | 4
Grade 3 Lung Infection-lung (Infections and infestations) | 15
Grade 5 Lung infection-lung (Infections and infestations) | 1
Grade 3 Lung infection-sinus (Infections and infestations) | 5
Grade 3 Lung infection-upper airway (Infections and infestations) | 1
Grade 3 Lung infection Unk ANC-bronchus (Infections and infestations) | 7
Grade 3 Lung infection Unk ANC-lung (Infections and infestations) | 6
Grade 3 Lung infection normal ANC-nose (Infections and infestations) | 1
Grade 3 Opportunistic infection associated w/lymphopenia (Infections and infestations) | 110
Grade 4 Opportunistic infection associated w/lymphopenia (Infections and infestations) | 1
Grade 5 Opportunistic infection associated w/lymphopenia (Infections and infestations) | 1
Grade 3 Viral hepatitis (Infections and infestations) | 1
Grade 5 Lung infection Unk ANC-bronchus (Infections and infestations) | 1
Grade 3 Skin infection Unk ANC-skin (Infections and infestations) | 1
Grade 3 Edema-head and neck (Blood and lymphatic system disorders) | 1
Grade 3 Edema-limb (Blood and lymphatic system disorders) | 9
Grade 3 Edema-trunk/genital (Blood and lymphatic system disorders) | 1
Grade 3 Lymphatics-other (Blood and lymphatic system disorders) | 3
Grade 3 Acidosis (Metabolism and nutrition disorders) | 3
Grade 3 Bicarbonate decrease (Metabolism and nutrition disorders) | 8
Grade 4 Bicarbonate decrease (Metabolism and nutrition disorders) | 8
Grade 3 GGT(Gamma-glutamyl transferase) (Metabolism and nutrition disorders) | 1
Grade 3 Hypercalcemia (Metabolism and nutrition disorders) | 1
Grade 4 Hypercalcemia (Metabolism and nutrition disorders) | 7
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 109
Grade 4 Hyperglycemia (Metabolism and nutrition disorders) | 14
Grade 3 Hyperkalemia (Metabolism and nutrition disorders) | 17
Grade 4 Hyperkalemia (Metabolism and nutrition disorders) | 6
Grade 3 Hypermagnesemia (Metabolism and nutrition disorders) | 7
Grade 4 Hypermagnesemia (Metabolism and nutrition disorders) | 1
Grade 3 Hypernatremia (Metabolism and nutrition disorders) | 2
Grade 3 Hypocalcemia (Metabolism and nutrition disorders) | 98
Grade 4 Hypocalcemia (Metabolism and nutrition disorders) | 20
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 120
Grade 4 Hypokalemia (Metabolism and nutrition disorders) | 15
Grade 3 Hypomagnesemia (Metabolism and nutrition disorders) | 5
Grade 4 Hypomagnesemia (Metabolism and nutrition disorders) | 2
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 186
Grade 4 Hyponatremia (Metabolism and nutrition disorders) | 10
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 236
Grade 4 Hypophosphatemia (Metabolism and nutrition disorders) | 11
Grade 3 Device/prosthesis (Musculoskeletal and connective tissue disorders) | 1
Grade 3 Fracture (Musculoskeletal and connective tissue disorders) | 8
Grade 3 Gait/walking (Musculoskeletal and connective tissue disorders) | 8
Grade 4 Gait/walking (Musculoskeletal and connective tissue disorders) | 1
Grade 3 Muscle weakness-lower extrem. (Musculoskeletal and connective tissue disorders) | 3
Grade 4 Muscle weakness-whole body (Musculoskeletal and connective tissue disorders) | 1
Grade 3 Muscle weakness-whole body (Musculoskeletal and connective tissue disorders) | 12
Grade 3 Musculoskeletal-other (Musculoskeletal and connective tissue disorders) | 5
Grade 3 Soft tissue-abdomen (Musculoskeletal and connective tissue disorders) | 1
Grade 3 Ataxia (Nervous system disorders) | 5
Grade 3 CNS ischemia (Nervous system disorders) | 1
Grade 4 CNS ischemia (Nervous system disorders) | 3
Grade 3 Confusion (Nervous system disorders) | 16
Grade 4 Confusion (Nervous system disorders) | 4
Grade 3 Dizziness (includes lightneadedness, disequilibrium & vertigo) (Nervous system disorders) | 29
Grade 4 Dizziness (includes lightheadedness, disequilibrium & vertigo) (Nervous system disorders) | 4
Grade 3 Encephalopathy (Nervous system disorders) | 1
Grade 3 Involuntary movement (Nervous system disorders) | 2
Grade 3 Irritability (Nervous system disorders) | 1
Grade 4 Memory impairment (Nervous system disorders) | 1
Grade 3 Mental status (Nervous system disorders) | 3
Grade 3 Mood alteration (agitation, anxiety, depression, euphoria) (Nervous system disorders) | 22
Grade 4 Mood alteration (agitation, anxiety, depression, euphoria) (Nervous system disorders) | 3
Grade 3 Mood/conscious change (Nervous system disorders) | 1
Grade 3 Neurology-other (Nervous system disorders) | 2
Grade 3 Neuropathy-motor (Nervous system disorders) | 71
Grade 4 Neuropathy-motor (Nervous system disorders) | 9
Grade 3 Psychosis (Nervous system disorders) | 3
Grade 3 Seizure (Nervous system disorders) | 3
Grade 3 Sensory Neuropathy (Nervous system disorders) | 73
Grade 4 Sensory neuropathy (Nervous system disorders) | 5
Grade 3 Somnolence (Nervous system disorders) | 8
Grade 4 Somnolence (Nervous system disorders) | 2
Grade 3 Syncope (Nervous system disorders) | 30
Grade 4 Syncope (Nervous system disorders) | 1
Grade 3 Tremor (Nervous system disorders) | 6
Grade 3 Weakness-motor neuropathy (Nervous system disorders) | 1
Grade 3 Blurred vision (Eye disorders) | 8
Grade 3 Cataract (Eye disorders) | 6
Grade 3 Flashing lights (Eye disorders) | 1
Grade 3 Ocular-other (Eye disorders) | 1
Grade 3 Photophobia (Eye disorders) | 1
Grade 3 Retinal detachment (Eye disorders) | 1
Grade 3 Abdomen NOS (General disorders) | 12
Grade 3 Anus (General disorders) | 1
Grade 3 Bone (General disorders) | 6
Grade 3 Buttock (General disorders) | 2
Grade 3 Cardiac/heart (General disorders) | 3
Grade 3 Chest/thorax NOS (General disorders) | 4
Grade 3 Chest wall (General disorders) | 2
Grade 3 Esophagus (General disorders) | 2
Grade 3 External ear (General disorders) | 1
Grade 3 Extremity/limb (General disorders) | 18
Grade 4 Extremity/limb (General disorders) | 1
Grade 3 Face (General disorders) | 1
Grade 3 Head/headache (General disorders) | 11
Grade 3 Hip-left (General disorders) | 4
Grade 3 Hip-right (General disorders) | 5
Grade 3 Joint (General disorders) | 5
Grade 4 Joint (General disorders) | 1
Grade 3 Kidney (General disorders) | 1
Grade 3 Lower back (General disorders) | 14
Grade 4 Lower back (General disorders) | 4
Grade 3 Middle back (General disorders) | 15
Grade 3 Muscle (General disorders) | 6
Grade 3 Neck (General disorders) | 6
Grade 3 Neuralgia/peripheral nerve (General disorders) | 2
Grade 3 Oral cavity (General disorders) | 2
Grade 3 Pain NOS (General disorders) | 12
Grade 3 Pleura (General disorders) | 2
Grade 3 Rectum (General disorders) | 1
Grade 3 Rib (General disorders) | 2
Grade 3 Sinus (General disorders) | 1
Grade 3 Skin (General disorders) | 1
Grade 3 Stomach (General disorders) | 5
Grade 3 Throat pharynx/larynx (General disorders) | 5
Grade 4 Throat pharynx/larynx (General disorders) | 1
Grade 3 Tumor pain (General disorders) | 2
Grade 4 Tumor pain (General disorders) | 1
Grade 3 Upper back (General disorders) | 26
Grade 4 Upper back (General disorders) | 3
Grade 4 ARDS (Respiratory, thoracic and mediastinal disorders) | 4
Grade 5 Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Cough (Respiratory, thoracic and mediastinal disorders) | 14
Grade 3 DLCO (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28
Grade 4 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 58
Grade 4 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Grade 5 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 22
Grade 4 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Grade 3 Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Grade 4 Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Prolonged intubation (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 12
Grade 3 Bladder spasms (Renal and urinary disorders) | 2
Grade 4 Bladder spasms (Renal and urinary disorders) | 1
Grade 3 Creatinine increase (Renal and urinary disorders) | 23
Grade 4 Creatinine increase (Renal and urinary disorders) | 10
Grade 3 GU fistula-bladder (Renal and urinary disorders) | 1
Grade 3 Incontinence-urinary (Renal and urinary disorders) | 9
Grade 3 Renal failure (Renal and urinary disorders) | 7
Grade 4 Renal failure (Renal and urinary disorders) | 5
Grade 3 Renal-other (Renal and urinary disorders) | 6
Grade 3 Urinary frequency/urgency (Renal and urinary disorders) | 13
Grade 3 Urinary retention (Renal and urinary disorders) | 1
Grade 3 Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Grade 4 Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Grade 3 Sexual-other (Reproductive system and breast disorders) | 1
Grade 3 HN Operative Injury-neck (Surgical and medical procedures) | 1
Grade 3 Muscle operative Injury-joint (Surgical and medical procedures) | 1
Grade 3 Operative Injury-other (Surgical and medical procedures) | 2
Grade 3 Thrombosis/embolism (Vascular disorders) | 48
Grade 4 Thrombosis/embolism (Vascular disorders) | 5
Grade 3 Thrombosis/embolism (vasc acc) (Vascular disorders) | 5
Grade 4 Thrombosis/embolism (vasc acc) (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=303)
Grade 1 Allergic reaction/hypersensitivity (Immune system disorders) | 69
Grade 2 Allergic reaction/hypersensitivity (Immune system disorders) | 27
Grade 1 Rhinitis (Immune system disorders) | 43
Grade 2 Rhinitis (Immune system disorders) | 19
Grade 1 Auditory/ear-other (Ear and labyrinth disorders) | 16
Grade 2 Hearing w/o monitoring program (Ear and labyrinth disorders) | 16
Grade 2 Tinnitus (Ear and labyrinth disorders) | 31
Grade 2 Anemia (Blood and lymphatic system disorders) | 112
Grade 1 Ventricular Arrythmia (Cardiac disorders) | 52
Grade 2 Ventricular Arrythmia (Cardiac disorders) | 58
Grade 1 Constitutional symptoms-other (General disorders) | 48
Grade 2 Constitutional symptoms-other (General disorders) | 17
Grade 2 Fatigue (lethargy, malaise, asthenia) (General disorders) | 84
Grade 1 Fever (absence of neutropenia) (General disorders) | 131
Grade 2 Fever (absence of neutropenia) (General disorders) | 82
Grade 1 Insomnia (General disorders) | 53
Grade 2 Insomnia (General disorders) | 26
Grade 1 Rigors/chills (General disorders) | 47
Grade 1 Sweating (General disorders) | 54
Grade 2 Sweating (General disorders) | 22
Grade 1 Weight loss (General disorders) | 17
Grade 1 Weight gain (General disorders) | 44
Grade 1 Alopecia (Skin and subcutaneous tissue disorders) | 22
Grade 2 Alopecia (Skin and subcutaneous tissue disorders) | 61
Grade 1 Dermatology-other (Skin and subcutaneous tissue disorders) | 38
Grade 2 Dermatology-other (Skin and subcutaneous tissue disorders) | 18
Grade 1 Dry skin (Skin and subcutaneous tissue disorders) | 50
Grade 2 Dry skin (Skin and subcutaneous tissue disorders) | 28
Grade 1 Flushing (Skin and subcutaneous tissue disorders) | 17
Grade 1 Pruritus (Skin and subcutaneous tissue disorders) | 18
Grade 1 Skin rash/desquamation (Skin and subcutaneous tissue disorders) | 100
Grade 2 Skin rash/desquamation (Skin and subcutaneous tissue disorders) | 82
Grade 1 Hot flashes (Endocrine disorders) | 15
Grade 2 Hypothyroidism (Endocrine disorders) | 22
Grade 1 Anorexia (Gastrointestinal disorders) | 27
Grade 2 Anorexia (Gastrointestinal disorders) | 133
Grade 1 Colitis (Gastrointestinal disorders) | 37
Grade 2 Colitis (Gastrointestinal disorders) | 35
Grade 1 Constipation (Gastrointestinal disorders) | 122
Grade 2 Constipation (Gastrointestinal disorders) | 107
Grade 1 Dehydration (Gastrointestinal disorders) | 15
Grade 2 Dehydration (Gastrointestinal disorders) | 30
Grade 1 Diarrhea (Gastrointestinal disorders) | 66
Grade 2 Diarrhea (Gastrointestinal disorders) | 111
Grade 1 Dry mouth (Gastrointestinal disorders) | 47
Grade 2 Dry mouth (Gastrointestinal disorders) | 21
Grade 1 Dysphagisa (Gastrointestinal disorders) | 33
Grade 2 Dysphagia (Gastrointestinal disorders) | 56
Grade 1 Esophagitis (Gastrointestinal disorders) | 23
Grade 2 Esophagitis (Gastrointestinal disorders) | 65
Grade 1 GI-other (Gastrointestinal disorders) | 33
Grade 1 Heartburn (Gastrointestinal disorders) | 34
Grade 1 Mucositis/Stomatitis (Gastrointestinal disorders) | 96
Grade 2 Mucositis/Stomatitis (Gastrointestinal disorders) | 60
Grade 1 Nausea (Gastrointestinal disorders) | 59
Grade 2 Nausea (Gastrointestinal disorders) | 149
Grade 1 Taste alteration (Gastrointestinal disorders) | 28
Grade 2 Taste alteration (Gastrointestinal disorders) | 14
Grade 1 Vomiting (Gastrointestinal disorders) | 68
Grade 2 Vomiting (Gastrointestinal disorders) | 108
Grade 1 Hemorrhage-lower GI (Blood and lymphatic system disorders) | 19
Grade 1 Alkaline phosphatase increase (Hepatobiliary disorders) | 181
Grade 2 Alkaline phosphatase increase (Hepatobiliary disorders) | 31
Grade 1 Bilirubin increase (Hepatobiliary disorders) | 78
Grade 2 Bilirubin increase (Hepatobiliary disorders) | 26
Grade 1 Hypoalbuminemia (Hepatobiliary disorders) | 40
Grade 2 Hypoalbuminemia (Hepatobiliary disorders) | 208
Grade 1 SGOT (AST) increase (Hepatobiliary disorders) | 171
Grade 2 SGOT (AST) increase (Hepatobiliary disorders) | 28
Grade 1 SGPT (ALT) increase (Hepatobiliary disorders) | 168
Grade 2 SGPT (ALT) increase (Hepatobiliary disorders) | 45
Grade 2 Opportunistic infection (Infections and infestations) | 20
Grade 2 Infection (documented clinically or microbiologically) (Infections and infestations) | 26
Grade 1 Edema-head and neck (Blood and lymphatic system disorders) | 23
Grade 1 Edema-limb (Blood and lymphatic system disorders) | 118
Grade 2 Edema-limb (Blood and lymphatic system disorders) | 36
Grade 1 Lymphatics-other (Blood and lymphatic system disorders) | 16
Grade 1 Bicarbonate decrease (Metabolism and nutrition disorders) | 219
Grade 2 Bicarbonate decrease (Metabolism and nutrition disorders) | 34
Grade 1 Hypercalcemia (Metabolism and nutrition disorders) | 32
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 15
Grade 2 Hyperglycemia (Metabolism and nutrition disorders) | 165
Grade 1 Hyperkalemia (Metabolism and nutrition disorders) | 95
Grade 2 Hyperkalemia (Metabolism and nutrition disorders) | 34
Grade 1 Hypermagnesemia (Metabolism and nutrition disorders) | 31
Grade 1 Hypernatremia (Metabolism and nutrition disorders) | 49
Grade 2 Hypocalcemia (Metabolism and nutrition disorders) | 151
Grade 1 Hypokalemia (Metabolism and nutrition disorders) | 162
Grade 1 Hypomagnesemia (Metabolism and nutrition disorders) | 75
Grade 2 Hypomagnesemia (Metabolism and nutrition disorders) | 36
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 104
Grade 2 Hypophosphatemia (Metabolism and nutrition disorders) | 54
Grade 1 Gait/walking (Musculoskeletal and connective tissue disorders) | 18
Grade 1 Joint-function (Musculoskeletal and connective tissue disorders) | 15
Grade 1 Muscle weakness-whole body (Musculoskeletal and connective tissue disorders) | 35
Grade 2 Muscle weakness-whole body (Musculoskeletal and connective tissue disorders) | 29
Grade 1 Musculoskeletal-other (Musculoskeletal and connective tissue disorders) | 46
Grade 1 Confusion (Nervous system disorders) | 66
Grade 2 Confusion (Musculoskeletal and connective tissue disorders) | 26
Grade 1 Dizziness (Nervous system disorders) | 96
Grade 2 Dizziness (Nervous system disorders) | 72
Grade 1 Memory impairment (Nervous system disorders) | 22
Grade 2 Memory impairment (Nervous system disorders) | 14
Grade 1 Mood alteration (Nervous system disorders) | 99
Grade 2 Mood alteration (Nervous system disorders) | 97
Grade 1 Neurology-other (Nervous system disorders) | 16
Grade 1 Neuropathy-motor (Nervous system disorders) | 74
Grade 2 Neuropathy-motor (Nervous system disorders) | 84
Grade 1 Sensory -neuropathy (Nervous system disorders) | 77
Grade 2 Sensory-neuropathy (Nervous system disorders) | 118
Grade 2 Somnolence (Nervous system disorders) | 28
Grade 1 Tremor (Nervous system disorders) | 56
Grade 2 Tremor (Nervous system disorders) | 27
Grade 1 Blurred vision (Eye disorders) | 146
Grade 2 Blurred vision (Eye disorders) | 32
Grade 1 Ocular-other (Eye disorders) | 24
Grade 1 Abdomen (General disorders) | 31
Grade 2 Bone (General disorders) | 16
Grade 1 Chest-thorax (General disorders) | 16
Grade 1 Chest wall (General disorders) | 16
Grade 1 Extremity-limb (General disorders) | 36
Grade 2 Extremity-limb (General disorders) | 42
Grade 1 Head-headache (General disorders) | 51
Grade 2 Head-headache (General disorders) | 25
Grade 2 Hip-left (General disorders) | 16
Grade 1 Joint (General disorders) | 29
Grade 2 Joint (General disorders) | 23
Grade 1 Lower back (General disorders) | 35
Grade 2 Lower back (General disorders) | 57
Grade 1 Middle back (General disorders) | 32
Grade 2 Middle back (General disorders) | 24
Grade 1 Muscle (General disorders) | 18
Grade 1 Neck (General disorders) | 17
Grade 1 Pain NOS (General disorders) | 48
Grade 2 Pain NOS (General disorders) | 27
Grade 1 Stomach (General disorders) | 23
Grade 1 Throat pharynx-larynx (General disorders) | 15
Grade 1 Upper back (General disorders) | 57
Grade 2 Upper back (General disorders) | 76
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 158
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 72
Grade 1 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 46
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28
Grade 1 Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 23
Grade 2 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 66
Grade 1 Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 19
Grade 2 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20
Grade 1 Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 30
Grade 2 Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 17
Grade 1 Creatinine increase (Renal and urinary disorders) | 112
Grade 2 Creatinine increase (Renal and urinary disorders) | 62
Grade 1 Incontinence-urinary (Renal and urinary disorders) | 27
Grade 2 Incontinence-urinary (Renal and urinary disorders) | 17
Grade 1 Renal-other (Renal and urinary disorders) | 23
Grade 1 Urinary frequency-urgency (Renal and urinary disorders) | 75
Grade 2 Urinary frequency-urgency (Renal and urinary disorders) | 27
Grade 2 Thrombosis/embolism (Vascular disorders) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No